CLINICAL TRIAL: NCT07183254
Title: Resting-state Functional Imaging in Chronic Consumption of Non-energetic Artificial Sweeteners
Brief Title: Resting-state Imaging and Chronic Consumption of Non-Nutritive SweetenerS
Acronym: RNSS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RBHP 2025 PICKERING
Record Dates: First submitted 2025-09-08; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers - Male and Female
Keywords: non-nutritive sweeteners; non- and low consumers; high consumers; resting-state MRI; diffusion tensor imaging (DTI); reward circuit; resting-state functional connectivity
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Intervention Model Description: Two Groups:
  * Healthy subjects, both low and non-sweetener consumers (~ 8 mg ± 5,05 mg / day), will have to consume 660 ml of sweetened beverage (2 cans) per day, which corresponds to an estimate of more than 87 mg of a mixture of acesulfame K and aspartame, for 5 weeks.
  * Healthy subjects, high sweetener consumers (~80 mg ± 91,72 mg / day)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects with low or no sweetener consumption, with a gender ratio close to 50/50 (Experimental): Subjects will be included:
  * Men and women aged 18 to 30 (and in good health)
  * Having low or no sweetener consumption (~8 mg ± 5.05 mg/day)
  * Having a BMI of 18.5 < 24.9
  * For young women: having effective contraception maintained throughout the study
  * Able to give informed consent to participate in the research
  * Affiliation to a Social Security scheme
  Interventions: Other: administration of questionnaires; Other: carrying out a MRI scan; Dietary Supplement: Can distribution visit for subjects in the "non/low" sweetener consumption group
- Subjects with high sweetener consumption, with a gender ratio close to 50/50 (Experimental): Subjects will be included:
  * Men and women aged 18 to 30 (and in good health)
  * Having high sweetener consumption (~80 mg ± 91.72 mg/day)
  * Having a BMI of 18.5 < 24.9
  * For young women: having effective contraception maintained throughout the study
  * Able to give informed consent to participate in the research
  * Affiliation to a Social Security scheme
  Interventions: Other: administration of questionnaires; Other: carrying out a MRI scan

INTERVENTIONS:
Other: administration of questionnaires — During this visit, the investigator will again explain the study objectives and procedure. Once these explanations have been provided, healthy volunteers will be able to give their informed consent to participate.
  After signing the consent form, the following will be conducted during this visit:
  * A medical examination.
  * An electronic questionnaire including two consumption frequency assessment tools, adapted in French, to measure daily sugar and artificial sweetener intake.
  * Five tests assess the level of dependence on alcohol, drugs (cannabis, solvents, tranquilizers, barbiturates, cocaine, stimulants, hallucinogens, or narcotics), gambling, video games, and possible eating disorders. Volunteers with a score deemed above the norm for at least one of these six tests will be excluded from this study.
  * A urine screening test for drug use (cannabis, opiates, amphetamines, cannabinoids, benzodiazepines, cocaine) will be performed during this visit.
  Other Names: Visit 1
Other: carrying out a MRI scan — A functional exploration using resting-state fMRI and microstructural tissue organization using DTI will take place in the days following the inclusion visit, depending on the availability of "research" slots in the Department of Radiology and Imaging, Clermont-Ferrand University Hospital.
  Other Names: Visit 2 - Resting-state fMRI and DTI - Department of Radiology and Imaging
Dietary Supplement: Can distribution visit for subjects in the "non/low" sweetener consumption group — During this visit, scheduled following the MRI, subjects will go to the PIC/CIC where they will be given cans for the 5 weeks of the nutritional intervention (660 ml of sweetened beverage, or 2 cans per day). Subjects will be advised to arrive by car if possible and to park in the PIC/CIC parking lot at the foot of the building. Drinks will be provided to the subject in one or two batches (with an additional visit to the center to pick up any missing drinks) at the subject's convenience. They will also receive instructions for completing the electronic questionnaire to assess daily sugar and sweetener consumption. Subjects will complete this questionnaire weekly, which they will receive by email. Their email address will be collected during this visit.
  Other Names: Visit 3
  Arms: Subjects with low or no sweetener consumption, with a gender ratio close to 50/50
Other: carrying out a MRI scan — A functional exploration using resting-state fMRI and microstructural tissue organization using DTI, post-nutritional intervention (5 weeks) in non- and low-sugar consumers: this exploration will take place depending on the availability of "research" slots at the Department of Radiology and Imaging, Clermont-Ferrand University Hospital.
  Other Names: Visit 4
  Arms: Subjects with low or no sweetener consumption, with a gender ratio close to 50/50

SUMMARY:
Non-nutritive sweeteners are used as a substitute for simple sugars to improve the palatability of food products without increasing their sugar and calorie content. They represent a global market of 7 billion euros, with an annual growth of 5%. Reducing their consumption therefore seems to be excluded. Some studies have focused on the impacts of these substances on brain activity. According to a recent study, continuous consumption of low doses of saccharin in adult mice significantly decreases the level of dopamine in the prefrontal cortex and significantly increases striatal dopamine, which modifies decision-making strategies. Resting-state functional Magnetic Resonance Imaging (r-fMRI) studies in humans have also shown that an increase in striatal dopaminergic activity modifies the resting-state functional connectivity of brain regions linked to the reward circuit. r-fMRI allows the characterization of brain networks and the strength of correlations between brain regions, without any specific task being required. It is a rapid, non-invasive technique that can measure changes in brain functional connectivity.

In addition to r-fMRI, diffusion tensor imaging (DTI) is able to assess white matter microstructure and the integrity or otherwise of fiber tracts. Several parameters such as the fractional anisotropy (FA), coefficient of white matter, mean diffusivity, and radial diffusivity can be modified in the event of changes in functional connectivity, reflecting axonal rearrangements, not visible on conventional MRI sequences. Based on previous research, investigators hypothesize that (1) chronic consumption of non-nutritive artificial sweeteners increases striatal dopaminergic activity. (2) This modification is accompanied by changes in resting-state functional connectivity in brain regions of interest associated with the reward circuit in healthy young adults.

Then, the primary objective of this study is to compare, in the resting state, the differences in functional connectivity of brain regions of interest between "non/low consumers" and "high consumers" of sweeteners at the start of the study using r-fMRI.

The key secondary objective of this study is to assess changes in brain connectivity using r-fMRI in non- and low-consuming subjects before and after a transient increase in their sweetener consumption over 5 weeks.

The secondary objectives include assessing daily sugar consumption (5-week follow-up), daily consumption of non-energy-rich artificial sweeteners (5-week follow-up), Body Mass Index (BMI), physical activity level, and white matter microstructure and fibrous tract integrity using a diffusion-weighted MRI (DTI) sequence.

DETAILED DESCRIPTION:
A single-center interventional study in 35 non- and low-consumers (approximately 8 mg/day) and 35 high-consumers (approximately 70 mg/day) selected, among other things, using a quantitative consumption frequency questionnaire on daily sugar and sweetener intake, whose frequency scale has been validated by a previous study.

The subjects recruited are healthy young adults, aged 18 to 30 years. An initial f-rMRI and DTI session will be performed for both groups (non- and low-consumers and high-consumers of sweeteners).

Then, a second session will be conducted after 5 weeks of nutritional intervention only in non- and low-consumers of sweeteners. During this period, subjects will be asked to consume 660 ml of sweetened carbonated beverages, the equivalent of 2 cans per day, with or without meals. They will also be asked to record their daily sugar and sweetener consumption, using an adapted version of the previously mentioned consumption frequency questionnaire, during this same period.

The study will observe initial differences in brain connectivity between non- and low-consumers and high-consumers of sweeteners, as well as changes in connectivity in non- and low-consumers before and after the nutritional intervention.

Comparison of functional connectivity between non- and low consumers and high consumers, as well as the change in connectivity before and after nutritional intervention in non- and low consumers will be performed by comparing connectivity matrices among all possible pairs of regions of interest, with a t-test for independent samples (between non- and low consumers and high consumers at t = 0) and dependent samples (non- and low consumers pre- and post-nutrition intervention; t = 0 and t = 5 weeks). Results will be expressed in terms of effect sizes and 95% confidence intervals.

At baseline (t = 0), the assessment of daily intake of simple sugars and BMI, as well as the level of physical activity, will be analyzed in relation to the consumption of non-nutritive artificial sweeteners, using a one-way ANOVA or a Kruskal-Wallis test, and a Chi-square test or a Fisher's exact test, respectively.

The assessment of intakes of simple sugars and non-nutritive artificial sweeteners during the 5 weeks of nutritional intervention (t = 5 weeks) in non- and low-consumers will be compared to the intakes of sugars and sweeteners estimated at t = 0, using a dependent-samples t-test or a Mann-Whitney test, if the conditions for applying the t-test are not met. The results will be expressed in terms of effect size and 95% confidence interval. To describe changes in white matter microstructure in non- and low-drinkers compared with high-drinkers, anisotropic fraction and ADC will be compared by Student's t-test or Mann-Whitney test. Results will be expressed as effect sizes and 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 30 (and in good health)
* Having low or no sweetener consumption (~8 mg ± 5.05 mg/day) or high consumption (~80 mg ± 91.72 mg/day)
* Having a BMI of 18.5 < 24.9
* For young women: having effective contraception maintained throughout the study
* Able to give informed consent to participate in the research
* Affiliation to a Social Security scheme

Exclusion Criteria:

* Refusing to participate in the research
* With impaired understanding, according to the investigator
* Volunteer under guardianship/curatorship/deprived of liberty or under legal protection
* Incompatibility of healthy volunteers with the medical imaging center's safety criteria for conducting 3 Tesla MRI experiments
* Presenting "contraindications" to an MRI examination without injection: presence of metal parts in the body (electronic devices such as a pacemaker, a neurostimulator, cochlear implant, prostheses, intraocular foreign bodies, etc.), claustrophobia, obesity
* Refusal to be informed in the event of an incidental discovery of an abnormality on MRI
* Volunteer with neurological disease, psychiatric or behavioral disorders*
* Volunteer with addiction*:

  * Nicotine: smoker or former smoker of less than 12 months;
  * Alcoholism - "AUDIT" test: Female score ≥ 6 and male score ≥ 7;
  * Drugs - "DAST-10": Score ≥ 1;
  * Gambling - "ICJE": Score ≥ 3
  * Video games - Modified DSM IV Video Game Addiction Test: More than 4 positive responses. - Positive urine drug screen
* Volunteer with an eating disorder (ED)*:

  o Eating disorder - "SCOFF": At least two positive responses. - Volunteers with at least one chronic condition (obesity, diabetes, cardiovascular, renal, or hepatic diseases, etc.)*
* Pregnant or breastfeeding women, or healthy subjects wishing to conceive during the current study year*
* Any illness, health condition, or history deemed incompatible with the trial by the investigator
* Volunteers following a specific or highly restrictive diet (vegetarians, vegans, or vegans; multiple dietary exclusions related to religion, food allergies or intolerances; diets related to intensive exercise or weight-loss)*
* Currently excluded from another study
* Currently participating in another clinical trial, or in the exclusion period, or having received a total compensation amount exceeding €6,000 in the 12 months preceding the start of the trial,

  * This study is part of a larger research project, also involving cognitive tasks and the measurement of food preferences. These exclusion criteria were therefore added in order to standardize the profile of the participants.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
1. At rest, functional connectivity between brain areas in healthy subjects, non/low consumers and high consumers of sweetener | High sweetner consumers: within 4 weeks after enrollment. Low or no sweetner consumer: within 4 weeks after enrollment and immediately after completion of the 5-weeks nutritional intervention.
  Resting-state functional magnetic resonance imaging (rs-fMRI) is a method that studies the connectivity of different regions of the nervous system. Based on the acquisition of the BOLD (Bond Oxygen Level Dependent) signal, this method focuses more specifically on the study of low-frequency fluctuations (<0.1 Hz) of this signal. The goal of resting-state imaging is to identify the synchronous activation of different regions of the brain and brainstem, in the absence of a stimulus or a task being performed. This activation can be observed between physically connected regions, or not, and demonstrates the involvement of these regions in a common network called the "Resting State Network" (RSN), which brings together different brain regions involved in common functions; this is referred to as "functional connectivity" between these regions. Areas of interest involved in the reward circuit (amygdala, nucleus accumbens, anterior insula, striatum, the prefrontal cortex, hypothalamus).

SECONDARY OUTCOMES:
Functional connectivity, at rest, before and after nutritional intervention in non- and low-sugar consumers (criterion for the key secondary objective). | Immediately after completion of the 5-weeks nutritional intervention.
  rs-fMRI
The amount of sugar consumed per day during the 5 weeks of nutritional intervention in non- and low-sugar consumers (mg/day). | Daily during the 5 weeks of the nutritional intervention among non-users and low consumers of sweeteners.
  Non-Nutritive Sweetener Food Frequency Questionnaire
The amount of artificial sweeteners consumed per day during the 5 weeks of nutritional intervention in non- and low-sugar consumers. (mg/day). | Daily during the 5 weeks of nutritional intervention in non- and low-sugar consumers.
  Non-Nutritive Sweetener Food Frequency Questionnaire
Body Mass Index (BMI) | At enrollment
  Body mass index (BMI) is a medical screening tool that measures the ratio of your height to your weight to estimate the amount of body fat you have. Healthcare providers calculate BMI by using weight in kilograms (kg) divided by the square of height in meters (m2). Healthy BMI range: 18.5 - 24.9
Level of physical activity (number of hours of exercise per week). | At enrollment
  Questionnaire.
  Physical activity will be categorized based on the number of hours of exercise per week as follows:
  * Low (< 2 hours/week)
  * Moderate (2-4 hours/week)
  * High (> 4 hours/week
The various tractography parameter characterizing the microstructure of the white matter: FA (fractional anisotropy), in brain regions in reward system. | High sweetner consumers: within 4 weeks after enrollment. Low or no sweetner consumer: within 4 weeks after enrollment and immediately after completion of the 5-weeks nutritional intervention.
  A medical image analysis platform (https://www.olea-medical.com/fr/solutions) is used for the analysis of diffusion tensor imaging (DTI) MRI sequence data. DTI parameters were measured from regions of interest (ROI) on brain structures involved in the reward circuit include, among others, the amygdala, the nucleus accumbens, the anterior insula, the striatum, the prefrontal cortex, and the hypothalamus.
  FA is a normalized scalar index ranging between 0 (completely isotropic diffusion, equal in all directions, e.g., cerebrospinal fluid) and 1(highly anisotropic diffusion, in a single direction, e.g., intact and well-aligned axons).
The various tractography parameters characterizing the microstructure of the white matter: diffusion parameters (axial and radial diffusion) in brain regions in reward system. | High sweetner consumers: within 4 weeks after enrollment. Low or no sweetner consumer: within 4 weeks after enrollment and immediately after completion of the 5-weeks nutritional intervention.
  A medical image analysis platform (https://www.olea-medical.com/fr/solutions) is used for the analysis of diffusion tensor imaging (DTI) MRI sequence data. DTI parameters were measured from regions of interest (ROI) on brain structures involved in the reward circuit include, among others, the amygdala, the nucleus accumbens, the anterior insula, the striatum, the prefrontal cortex, and the hypothalamus.
  Mean diffusivity (MD), Axial diffusivity (AD, diffusion along the principal axis of the nerve fibers) and radial diffusivity (RD, diffusion across the principal axis of the nerve fibers) in diffusion tensor imaging (DTI) are expressed in mm²/s, often reported as ×10-³ mm²/s.
  In normal white matter, MD is around 0.7-0.9 ×10-³ mm²/s, AD is approximately 1.1-1.3 ×10-³ mm²/s and RD is approximately 0.6-0.8 ×10-³ mm²/s.
The various tractography parameter characterizing the microstructure of the white matter: ADC (apparent diffusion coefficient) in brain regions in reward system. | High sweetner consumers: within 4 weeks after enrollment. Low or no sweetner consumer: within 4 weeks after enrollment and immediately after completion of the 5-weeks nutritional intervention.
  A medical image analysis platform (https://www.olea-medical.com/fr/solutions) is used for the analysis of diffusion tensor imaging (DTI) MRI sequence data. DTI parameters were measured from regions of interest (ROI) on brain structures involved in the reward circuit include, among others, the amygdala, the nucleus accumbens, the anterior insula, the striatum, the prefrontal cortex, and the hypothalamus.
  The ADC reflects the mean diffusivity of water within a voxel, accounting for both Brownian motion and tissue microstructural properties. It is reported in ×10-³ mm²/s, with normal values of ~0.7-0.9 in white matter, ~0.8-1.0 in gray matter, and ~3.0 in cerebrospinal fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle Pickering, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No